CLINICAL TRIAL: NCT02443857
Title: Feasibility of a New Pediatric Arm Rehabilitation Robot ChARMin: A Monocentric Interventional Study
Brief Title: Feasibility of a New Pediatric Arm Rehabilitation Robot ChARMin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huub van Hedel (Other)
Responsible Party: Sponsor-Investigator, Huub van Hedel, Head of Research and Therapies Rehabilitation Center for Children and Adolescents, University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ChARMin
Record Dates: First submitted 2015-04-16; First posted 2015-05-14 (Estimated); Last update posted 2025-03-11 (Actual); Status verified 2024-12

CONDITIONS: Nervous System Diseases
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ChARMin (Experimental): Single-arm only
  Interventions: Device: ChARMin

INTERVENTIONS:
Device: ChARMin — The aim is to investigate the applicability (technical aspects, patient-related aspects, operability/handling of the robot, the different control modes of the device, safety and the software interface) of ChARMin.
  Other Names: ChARMin-1
Device: ChARMin — The aim is to determine whether differences between game scores, kinematic and kinetic metrics provided by ChARMin, additionally applied physiological measures and adverse events differ when participants train with the free non-supported mode, the assist-as-needed mode and the fully guided mode.
  Other Names: ChARMin-2
Device: ChARMin — The aim is to determine the psychometric properties (validity, reliability and responsiveness) of the assessments integrated in ChARMin.
  Other Names: ChARMin-3
Device: ChARMin — The aim is to describe the application of the system in 30 participants and evaluate the concomitant changes in upper extremity motor function (open labelled interventional study without control group).
  Other Names: ChARMin-4
Device: ChARMin — The aim is to perform specific motor learning studies in 120 patients investigating whether children with neurological diagnoses can improve arm and hand task performance during repetitive training with ChARMin, are able to retain improved levels of task performance and how task performance is influenced by other interventions.
  Other Names: ChARMin-5
Device: ChARMin — The aim is to perform an ecological study monitoring safety, functional progress and (changes in) the application of ChARMin in 120 participants following an in- or out-patient program (comparable to subproject ChARMin-4).
  Other Names: ChARMin-6

SUMMARY:
The purpose of this study is to investigate the applicability and feasibility of the newly developed robot platform for upper extremity therapy ("ChARMin") in children undergoing neurorehabilitation.

DETAILED DESCRIPTION:
Background and Rationale: Children with neurological diagnoses including congenital or acquired brain lesions often have impaired upper extremity function that limits activities of daily life and independence. While several rehabilitation technologies in the clinical routines are being applied to improve upper extremity functions in these patients, the technology to train more severely affected children was not available so far. Since 3 years, the investigators are working together with the Sensory-Motor Systems Lab at ETH Zurich on a new robot platform specifically developed for upper extremity therapy in children (the 'Children's Arm Rehabilitation Mechatronic Interface' or 'ChARMin'). This group showed recently in a single blinded RCT that their adult upper extremity robot ARMin is an effective neurorehabilitation tool for adults after stroke (especially for the more severely affected patients). Now, that ChARMin is finished the investigators would like to study whether it is feasible to apply this prototype to children and adolescents undergoing neurorehabilitation.

Objective(s): As ChARMin was specifically developed for children and adolescents, the investigators first want to explore whether it is feasible to apply it to children and adolescents undergoing neurorehabilitation. Six studies will be performed with the following main objectives: (i) to investigate the applicability (technical aspects, patient-related aspects, operability/handling of the robot, the different control modes of the device, safety and the software interface) of ChARMin; (ii) to determine whether differences between game scores, kinematic and kinetic metrics provided by ChARMin, additionally applied physiological measures and adverse events differ when participants train with the free non-supported mode, the assist-as-needed mode and the fully guided mode; (iii) to determine the psychometric properties (validity, reliability and responsiveness) of the assessments integrated in ChARMin; (iv) to describe the application of the system in 30 participants and evaluate the concomitant changes in upper extremity motor function (open labelled interventional study without control group); (v) specific motor learning studies in 120 patients investigating whether children with neurological diagnoses can improve arm and hand task performance during repetitive training with ChARMin, are able to retain improved levels of task performance and how task performance is influenced by other interventions; (vi) to perform an ecological study monitoring safety, functional progress and (changes in) the application of ChARMin in 120 participants following an in- or out-patient program (comparable to subproject iv).

Outcome(s): The outcomes are in line with the objectives of each subproject. Some outcome measures are specifically performed for this study (e.g. safety, game scores, assessments integrated in ChARMin), others are clinically routinely applied measures (no additional burden for the patient). The investigators do not apply any invasive tools and assure that the amount of additional assessments will be limited to keep the burden for the participants acceptable.

Study design: Most projects are open labelled interventional studies investigating the applicability, safety and usability of a newly developed upper extremity robot ChARMin. Project (i) will investigate the feasibility of ChARMin in 30 children and adolescents. Project (ii) will be a randomized study investigating differences in the various measures between the 3 control modes of ChARMin. Project (iii) include psychometric studies where a single measurement is necessary (validity), or two repeated measurements are performed (within 3-7 days to determine reliability and between onset and end of rehabilitation to determine responsiveness). Project (v) consists of motor learning studies where a large number of repetitions are performed in a relative short time to determine changes in task performance, retention and generalizability. Projects (iv) and (vi) are open labelled interventional studies investigating the application of ChARMin and concomitant changes in upper extremity function without control group.

Measurements and procedures: Participants will be positioned in a comfortable position on a chair. After the required anthropometrics have been assessed, the ChARMin is adjusted and the cuffs of ChARMin will be fixated to the patient. Depending on the study, the participant will be informed and instructed what task/assessment or game will be made and what the goal is. Then, the participant will perform the task, while the investigator/therapist will be there to answer any questions, make sure the patient is comfortable, and to control the device, including the emergency buttons. Afterwards, the investigator/therapist will loosen the cuffs and assist if needed the participant getting out of the chair. The therapist will control the participant's skin and will ask for any other signs of discomfort. The duration of a session will remain within 45 minutes. In other sessions, clinical routine assessments will be performed.

Study Product / Intervention: The Children's Arm Rehabilitation Mechatronic Interface (ChARMin) is a newly developed upper extremity exoskeleton robot which can assist single joint movements and complex spatial reaching movements involving movements for shoulder, elbow, wrist and hand. As several subprojects are performed, the intervention could last a single training session of about 45 minutes, two or three sessions (for example to investigate reliability of assessments) or a longer training duration as prescribed by the medical doctor (e.g. for several weeks 3-5 times per week, as part of an intense a rehabilitation program).

Control Intervention (if applicable): NA (subproject 2: each child is its own control)

Number of Participants with Rationale: In general, the investigators plan to include about 30 participants per project as this number would results in a more or less normal distribution, and for psychometric studies, this is the number of participants needed to score a psychometric study of sufficient quality to be included in a best evidence synthesis.

Subproject (i): 30 participants. Subproject (ii): 30 participants. For subproject (iii) the investigators plan to recruit 60 participants (with at least 2 measurements per participant). Likely, the number might be smaller if participants agree to undergo 3 assessment sessions (first for validity, second for reliability and a final one for responsiveness). Reference values will be obtained in 40 healthy participants.

Subproject (iv): 30 participants. Subproject (v): Pilot motor learning studies will be performed in 40 participants, while the definite motor learning studies will be performed in 80 participants.

Subproject (vi): 120 participants. Please note, participants will likely contribute to more than 1 subproject with no high burden. Therefore, the total number of patients will therefore likely be smaller than 390.

Study Duration: 5 years

Study Schedule: Month Year of First-Participant-In (Mai 2015). Month Year of Last-Participant-Out (April 2020)

Study Centre(s): Monocentric study: Rehabilitation Center Affoltern am Albis

Statistical Considerations: The investigators will mainly report descriptive statistics. Normal distribution will be determined with the Shapiro-Wilk test. Comparisons between two dependent groups will be performed with Wilcoxon's or paired-t-test. Comparisons between two independent groups will be performed with a Mann-Whitney U test or a Student's t-test. Differences between three groups will be determined with a Friedman's test (dependent groups) or an ANOVA (independent groups). Relationships will be analysed with a Spearman's or Pearson correlation coefficient. Motor learning will be quantified with various measures: learning or adaptive rate will be fitted with a power or exponential regression; ratios will be calculated to quantify the transfer or retention between blocks of trials and retention.

GCP Statement: This study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki, the ICH-GCP or ISO EN 14155 (as far as applicable) as well as all national legal and regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 and 21 years
* Neurological diagnoses
* Impairment of the upper extremity (for projects (i) and (ii) we might also include patients without upper extremity impairments to cover a wide range of patients with different abilities)
* Other (non-neurological) diagnoses, who require intense training of the upper extremity

Exclusion Criteria:

* Strong adipositas, which makes it not possible to adjust the cuffs and orthoses to the anthropometrics of the participant
* Fixed contractures of the upper extremity that should be positioned in ChARMin
* Instabilities of bones or joints, fractures or osteoporosis/osteopenia
* Allergy against material of cuffs
* Open skin lesions of the upper extremity that should be positioned in ChARMin
* Luxations or subluxations of joints of the upper extremity that should be positioned in ChARMin
* Strong pain that increases while training in ChARMin*
* Injuries or lesioned nerves of the upper extremity that should be positioned in ChARMin*
* Strong spontaneous movements like ataxia, dyskinesia, myoclonus*
* Instable vital functions like pulmonal or cardiovascular conditions
* Implanted pace maker, defibrillator of the heart
* Implanted shunt by hydrocephalus*
* Implanted cochlear or baha*
* Uncooperative or aggressive behaviour
* Known or suspected non-compliance
* Severe cognitive deficits
* Inability to signal pain or discomfort
* Apraxia*
* Severe visual impairment (inability to see the screen)
* Severe spasticity (Ashworth 4)
* Severe epilepsy*
* Insufficient head stability
* Infections requiring isolation of the patient Contraindications marked with an * are relative contraindications. Final approval needs to be obtained from the medical doctor.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 430 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
ChARMin-1: Score on the feasibility questionnaire [points] | Up to 8 weeks
  The feasibility questionnaire is a self-developed tool, which covers the following areas:
  * Technical aspects:
  * Patient-related aspects:
  * Safety
  * Interface/Games/Assessments
ChARMin-2: Game Scores [points] | up to 24 weeks
  To calculate the game scores of each game, several kinematic and kinetic measures are recorded and processed during the games (for instance number of collected items)
ChARMin-3: Assessment battery integrated into the ChARMin software [points] | Up to 24 weeks
  The assessment battery consists of:
  * Range of motion
  * Workspace measurement
  * Quality of movement during targeted movements
  * Isometric strength measurement
  * Resistance to passive movement of the arm (stiffness)
  * Accuracy of performing a circle movement in the frontal plane.
ChARMin-3: Change from baseline of the assessment battery integrated into the ChARMin software [delta points] | Twice within 3-7 days
  To assess the reliability of the assessment battery.
  The assessment battery consists of:
  * Range of motion
  * Workspace measurement
  * Quality of movement during targeted movements
  * Isometric strength measurement
  * Resistance to passive movement of the arm (stiffness)
  * Accuracy of performing a circle movement in the frontal plane.
ChARMin-3: Change from baseline of the assessment battery integrated into the ChARMin software | At onset and end of the hospital stay, which covers an expected average of 7 weeks
  To assess the responsiveness of the assessment battery.
  The assessment battery consists of:
  * Range of motion
  * Workspace measurement
  * Quality of movement during targeted movements
  * Isometric strength measurement
  * Resistance to passive movement of the arm (stiffness)
  * Accuracy of performing a circle movement in the frontal plane.
ChARMin-4 and ChARMin-6: Change from baseline in the Box and Block Test [delta of the number of blocks transferred] | At onset and end of hospital stay, which covers an expected average of 7 weeks
  Individuals are seated at a table, facing a rectangular box that is divided into two square compartments of equal dimension by means of a partition. 150, 2.5 cm, colored, wooden cubes or blocks are placed in one compartment or the other. The participant is instructed to move as many blocks as possible, one at a time, from one compartment to the other for a period of 60 seconds. To administer the test, the examiner is seated opposite the individual in order to observe test performance. The BBT is scored by counting the number of blocks carried over the partition from one compartment to the other during the one-minute trial period. Patient's hand must cross over the partition in order for a point to be given, and blocks that drop or bounce out of the second compartment onto the floor are still rewarded with a point.
ChARMin-5: Game scores [points] | up to 24 weeks
  To calculate the game scores of each game, several kinematic and kinetic measures are recorded and processed during the games (for instance number of collected items)

SECONDARY OUTCOMES:
ChARMin-2: Joint angle measures provided by ChARMin [degrees] | up to 24 weeks
ChARMin-2: Force measures provided by ChARMin [Newton] | up to 24 weeks
ChARMin-2: Amplitude of muscle activation [microVolt] | up to 24 weeks
  Measured by surface electromyography
ChARMin-2: Palmar skin conductance [microVolt] | up to 24 weeks
  Measured via sympathetic skin response as a surrogate of the parasympathetic nervous system
ChARMin-2: Heart rate [beats per minute] | up to 24 weeks
  Measured via chest belt to get an idea about the cardiovascular intensity of the training.
ChARMin-2: Adverse events [number and kind of events] | up to 24 weeks
ChARMin-2: Score on the motivational questionnaire [points] | up to 24 weeks
ChARMin-4 and ChARMin-6: Change from baseline in the score of the assessment battery integrated into the ChARMin software [delta points] | At onset and end of hospital stay, which covers an expected average of 7 weeks
  The assessment battery consists of:
  * Range of motion
  * Workspace measurement
  * Quality of movement during targeted movements
  * Isometric strength measurement
  * Resistance to passive movement of the arm (stiffness)
  * Accuracy of performing a circle movement in the frontal plane.
ChARMin-4 and ChARMin-6: Change from baseline in the Nine-hole Peg Test [delta seconds] | At onset and end of hospital stay, which covers an expected average of 7 weeks
ChARMin-4 and ChARMin-6: Change from baseline in the brain reorganization measured by transcranial magnetic stimulation [delta milliseconds] | At onset and end of hospital stay, which covers an expected average of 7 weeks
  Transcranial magnetic stimulation to investigate whether the corticospinal tract is ipsi- or contralaterally reorganised
ChARMin-4 and ChARMin-6: Change from baseline in strength of fingers and hand [delta Newton] | At onset and end of hospital stay, which covers an expected average of 7 weeks
  Measured by dynamometry.

CONTACTS AND LOCATIONS:
Overall Officials: Hubertus JA van Hedel, PhD, Principal Investigator — Rehabilitation Center for Children and Adolescents of the University Children's Hospital Zurich
Locations (1):
- Rehabilitation Center for Children and Adolescents of the University Children's Hospital Zurich, Affoltern am Albis, Switzerland

REFERENCES:
- [Derived] Graser JV, Prospero L, Liesch M, Keller U, van Hedel HJA. Test-retest reliability of upper limb robotic exoskeleton assessments in children and youths with brain lesions. Sci Rep. 2022 Oct 6;12(1):16685. doi: 10.1038/s41598-022-20588-8. PMID 36202825
- [Derived] Graser JV, Bastiaenen CHG, Gut A, Keller U, van Hedel HJA. Contextual interference in children with brain lesions: a pilot study investigating blocked vs. random practice order of an upper limb robotic exergame. Pilot Feasibility Stud. 2021 Jun 25;7(1):135. doi: 10.1186/s40814-021-00866-4. PMID 34172085
- [Derived] Graser JV, Bastiaenen CHG, Keller U, van Hedel HJA. Contextual interference in children with brain lesions: protocol of a pilot study investigating blocked vs. random practice order of an upper limb robotic exergame. Pilot Feasibility Stud. 2020 Oct 15;6:156. doi: 10.1186/s40814-020-00694-y. eCollection 2020. PMID 33072397